CLINICAL TRIAL: NCT06575296
Title: A Phase I Study of SNDX 5613 (Revumenib) as Post-Transplant Maintenance After Allogeneic Hematopoietic Cell Transplant in Patients With KMT2A-Rearranged or NPM1-Mutated Acute Leukemia
Brief Title: Revumenib for the Treatment of Acute Leukemia in Patients Post-Allogeneic Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23520; NCI-2024-06738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23520 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Leukemia; Acute Leukemia of Ambiguous Lineage; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Childhood Acute Leukemia; Childhood Acute Leukemia of Ambiguous Lineage; Childhood Acute Lymphoblastic Leukemia; Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; revumenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (revumenib) (Experimental): Starting 50-150 days after alloHCT, patients receive revumenib PO QD or every 12 hours on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow biopsy during screening and may undergo ECHO during screening and as clinically indicated. Patients also undergo bone marrow aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Revumenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Other: Electronic Health Record Review — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Revumenib — Given PO
  Other Names: Menin-Mixed Lineage Leukemia Protein-Protein Interaction Inhibitor SNDX-5613; Menin-MLL Inhibitor SNDX-5613; Menin-MLL Interaction Inhibitor SNDX-5613; SNDX 5613; SNDX-5613; SNDX5613

SUMMARY:
This phase I trial tests the safety, side effects, best dose and effectiveness of revumenib in treating patients with acute leukemia after allogeneic stem cell transplant. Revumenib is in a class of medications called menin inhibitors. Revumenib targets and binds to the protein menin, thereby preventing the interaction between menin and the mixed lineage leukemia protein. Disrupting this interaction prevents the activation of specific genes that fuel the development of leukemia cells and inhibits the survival, growth, and production of certain kinds of leukemia cells. Giving revumenib may be safe, tolerable, and/or effective in treating patients with acute leukemia after allogeneic stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of revumenib as maintenance therapy in patients with KMT2A rearranged or NPM1 mutated acute leukemia after undergoing allogeneic hematopoietic cell transplantation (alloHCT).

II. Determine the recommended phase 2 dose (RP2D) of revumenib as maintenance therapy in patients with KMT2A rearranged (KMT2Ar) or NPM1 mutated (NPM1m) acute leukemia after undergoing alloHCT.

SECONDARY OBJECTIVES:

I. Assess overall survival (OS), relapse free survival (RFS), cumulative incidence of relapse (CIR), and composite graft versus host disease (GVHD)-free, relapse-free survival (GRFS) at 1 and 2 years from first dose of revumenib.

II. Non-relapse mortality (NRM) at 100 days 1 and 2 years after first dose of revumenib.

III. Evaluate the rate and grading of acute GVHD at 180 days after alloHCT. IV. Evaluate the incidence and grading of chronic GVHD (cGVHD) at 1 and 2 years after first dose of revumenib.

V. Evaluate minimal residual disease (MRD) using quantitative polymerase chain reaction (PCR) (NPM1m) or ClonoSeq (B-acute lymphoblastic leukemia [B-ALL]).

VI. Evaluate MRD using flow cytometry. VII. Evaluate the feasibility of maintenance therapy.

EXPLORATORY OBJECTIVES:

I. Evaluate immune cell populations and immune reconstitution after maintenance therapy.

II. Evaluate the inflammatory cytokine profile and levels. III. Evaluate detection of residual NPM1m error-corrected sequencing. IV. Develop and evaluate a novel KMT2Ar assay in detecting residual disease. V. Evaluate quality of life.

OUTLINE: This is a dose-escalation study of revumenib followed by a dose-expansion study.

Starting 50-150 days after alloHCT, patients receive revumenib orally (PO) once daily (QD) or every 12 hours on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow biopsy during screening and may undergo echocardiography (ECHO) during screening and as clinically indicated. Patients also undergo bone marrow aspiration and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 2 years post-treatment start.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WHO ARE SCHEDULED TO UNDERGO HEMATOPOIETIC CELL TRANSPLANTATION (HCT) OR THOSE WHO HAVE UNDERGONE HCT: Documented informed consent of the participant and/or legally authorized representative
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Agreement to allow the use of archival tissue from diagnostic tumor biopsies; if unavailable, exceptions may be granted with study principal investigator (PI) approval
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Participant is willing and able to adhere to the study visit schedule and other protocol requirements
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Age: >= 2 years
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Have a date for transplant within the next 4 weeks or have received transplant within the last 4 months
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Participant was diagnosed with an acute leukemia as defined by the World Health Organization (WHO) 5th edition criteria for acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or acute leukemia with ambiguous lineage
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Participant must meet one of the following disease characteristics:

  * Confirmed NPM1m AML with at least one of the following additional characteristics

    * FLT3-ITD co-mutation
    * Pre-transplant MRD+ disease by flow cytometry or real time polymerase chain reaction (qPCR)
    * Requires more than one AML induction regimen to acquire complete response (CR)1
    * In second or later complete remission
  * Confirmed KMT2Ar acute leukemia obtained by fluorescence in situ hybridization (11q23 MLL-break apart fluorescence in situ hybridization [FISH]) or next-generation sequencing (NGS)
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Any donor (sibling, unrelated, mismatched related/unrelated, cord and haploidentical) or graft source (peripheral blood [PB] stem cell or bone marrow [BM]) will be included
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Conditioning regimen: investigator's choice based on center guidelines
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: GVHD prophylaxis: investigator's choice based on center guidelines
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Patients receiving menin inhibitors prior to alloHCT are eligible
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Negative serum pregnancy test for female patients of childbearing potential who have already undergone alloHCT
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: If a female of childbearing potential, must be willing to use a highly effective method of contraception or double barrier method from the time of enrollment through 120 days following the last study drug dose
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: If male of childbearing potential, must agree to use barrier contraception from the time of enrollment through 120 days following the last study drug dose

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Participant has an Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky Performance Status (KPS) >= 70, or a Lansky Performance Score of >= 70 (if aged < 18 years)
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Participant must be eligible for alloHCT by City of Hope (COH) standard operating procedure (SOP) guidelines
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Patients should be in complete remission (CR) by day + 30 (± 7 days) post-HCT BM biopsy
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: No evidence of active or uncontrolled infection at the time of start of revumenib therapy
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participant has an ECOG =< 2 or KPS >= 70, or Lansky Performance Score of >= 70 if aged < 18 years
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: No active grade 2-4 acute GVHD (prednisone dose of =< 0.5 mg/kg daily is allowed)
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Hemoglobin (Hgb) >= 9. Transfusion or growth factors are not allowed to achieve these levels
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Platelets >= 75 thousand (k). Transfusion or growth factors are not allowed to achieve these levels
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Patients must be fully engrafted after HCT, defined as absolute neutrophil count (ANC) >= 500 for 3 days. Patients may NOT be given granulocyte colony-stimulating factor (GCSF) to meet eligibility criteria; however, they may receive GCSF after start of treatment
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: No morphologic evidence of relapse post-HCT (pre-HCT MRD+ is)
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participant is between day + 50 and + 150 after first alloHCT with no morphologic evidence of relapse post-HCT
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless considered to be due to Gilbert's syndrome)

  * Note: Participants who are < 75 years of age may have a bilirubin of =< 3.0 x ULN. Patients with abnormal liver function tests (LFTs) in the context of active GVHD will not be included
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Aspartate aminotransferase (AST) =< 2.5 x ULN
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Alanine aminotransferase (ALT) =< 2.5 x ULN
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: QTc using Fridericia's correction (QTcF) =< 450 msec (males) or =< 470 msec (females)
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Ejection fraction (EF) of >= 50% by echocardiogram or multigated acquisition (MUGA) scan
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula

Exclusion Criteria:

* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Prior diagnosis of acute promyelocytic leukemia
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Participants who are unable to take a strong CYP3A4 inhibitor such as voriconazole or posaconazole. Note: Patients must be taking a strong CYP3A4 inhibiting antifungal at least 7 days prior to starting revumenib cycle 1
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Patients requiring the concurrent use of medications known or suspected to prolong the QT/corrected QT (QTc) interval, with the exception of drugs with low risk of QT/QTc prolongation that are used as standard supportive therapies (e.g., diphenhydramine, famotidine, ondansetron, bactrim, tacrolimus, azoles)
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: History of or any concurrent condition, therapy, laboratory abnormality, or allergy to excipients that in the investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate
* PATIENTS WHO ARE SCHEDULED TO UNDERGO HCT OR THOSE WHO HAVE UNDERGONE HCT: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Participant has detectable human immunodeficiency virus (HIV) viral load within the previous 6 months (must have viral load testing prior to study enrollment if participant has a known history of HIV 1/2 antibodies)
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Active uncontrolled hepatitis B or C, defined as hepatitis B or C virus (HBV/HCV) surface antigen positive and HBV/HCV core antibody positive, with positive HBV/HCV deoxyribonucleic acid (DNA), or HBV/HCV positive core antibody alone with positive HBV/HCV DNA
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Hepatitis C, defined as positive HCV antibody with reflex to positive HCV ribonucleic acid (RNA)
* PATIENTS WHO HAVE NOT YET UNDERGONE HCT: Other active malignancy; patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Active grade II-IV acute GVHD, chronic GVHD (moderate or severe) and/or requiring systemic steroids with prednisone dose equivalent of >= 0.25mg/kg within 4 weeks of revumenib administration
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participant has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participants who are unable to take a strong CYP3A4 inhibitor such as voriconazole or posaconazole. Note: Patients must be taking a strong CYP3A4 inhibiting antifungal at least 7 days prior to starting revumenib in cycle 1
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Patients requiring the concurrent use of medications known or suspected to prolong the QT/QTc interval, with the exception of drugs with low risk of QT/QTc prolongation that are used as standard supportive therapies (e.g., diphenhydramine, famotidine, ondansetron, bactrim, tacrolimus, and azoles)
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Female participant who is pregnant or lactating
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participant has a malabsorption syndrome or other condition that precludes enteral route of administration
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Participant has chronic respiratory disease that requires continuous oxygen, or significant renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect participation in this study
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Cardiac disease: any of the following within the 6 months prior to study entry:

  * Myocardial infarction
  * Uncontrolled/unstable angina
  * Congestive heart failure (New York Heart Association Classification class >= II)
  * Life-threatening or uncontrolled arrhythmia
  * Cerebrovascular accident
  * Transient ischemic attack
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: Gastrointestinal disease:

  * Any gastrointestinal issue of the upper gastrointestinal (GI) tract likely to affect oral drug absorption or ingestion (e.g., gastric bypass, gastroparesis, etc.)
  * Cirrhosis with a Child-Pugh score of B or C
* CRITERIA TO PROCEED TO MAINTENANCE THERAPY WITH REVUMENIB: GVHD: Signs or symptoms of acute or cGVHD > grade 0 within 4 weeks of enrollment. Patients may be on physiological doses of steroids

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-04-29 (Estimated); Study Completion 2028-04-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Start of protocol therapy up to 2 years
  Will evaluate toxicity as graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5, including dose limiting toxicity (DLT). The toxicity/adverse event information recorded on each subject will include type, severity, duration, and attribution/association with the study regimen and DLT occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limited to infections, other adverse events of special interest, and serious adverse events.

SECONDARY OUTCOMES:
Molecular response | Up to 2 years
  Will evaluate molecular response using quantitative polymerase chain reaction for NPM1 mutated acute myeloid leukemia and ClonoSeq for B-acute lymphoblastic leukemia, per standard of care.
Overall survival (OS) | Start of protocol therapy to death, assessed up to 2 years
  OS will be censored at last follow-up if patients are known to be alive. Survival endpoints will be analyzed using Kaplan-Meier curves.
Relapse free survival (RFS) | Start of protocol therapy to relapse/progression or death, assessed up to 2 years
  RFS will be censored at last follow-up if patients are alive and relapse/progression-free. Survival endpoints will be analyzed using Kaplan-Meier curves.
Graft versus host disease (GVHD)-free/relapse survival (GRFS) | Start of protocol therapy to first observation of developing grade 3-4 acute GVHD, chronic GVHD requiring systemic therapy, relapse/progression, or death, assessed up to 2 years
  GRFS will be censored at last follow-up if patients are known to be alive and free of any event of interest. Survival endpoints will be analyzed using Kaplan-Meier curves.
Cumulative incidence of relapse/progression | Start of protocol therapy to relapse/progression, assessed up to 2 years
  Death without relapse/progression is considered a competing risk. Surviving patients with no history of relapse/progression are censored at the time of last follow-up. Competing risks endpoints will be analyzed using the curves of cumulative incidence.
Cumulative incidence of non-relapse mortality (NRM) | Start of protocol therapy to death without relapse/progression, assessed up to 2 years
  Relapse/progression is considered a competing risk. Surviving patients with no history of relapse/progression are censored at the time of last follow-up. Competing risks endpoints will be analyzed using the curves of cumulative incidence.
Rate of acute GVHD | Up to 180 days post hematopoietic cell transplantation (HCT)
  Will evaluate rate of acute GVHD of grades 2-4 and 3-4 by day 180 post-HCT. Documented/biopsy proven acute GVHD is graded according to Mount Sinai Acute Graft Versus Host Disease International Consortium Grading System. Time to event is measured from date of transplant to first documented/biopsy proven acute GVHD onset date. Acute GVHD will be censored at the time of last follow-up if patients remain alive and free of relapse/progression.
Cumulative incidence of chronic GVHD | Start of protocol therapy to documented/biopsy proven chronic GVHD, assessed up to 2 years
  Will evaluate documented/biopsy proven chronic GVHD as scored according to National Institutes of Health Consensus Staging. Disease relapse/progression or NRM are considered competing risk events. Chronic GVHD will be censored at the time of last follow-up if patients remain alive and free of relapse/progression. Competing risks endpoints will be analyzed using the curves of cumulative incidence.
Ability to complete at least 7 cycles of revumenib therapy | Up to 2 years
  Feasibility will be defined as ability to complete at least 7 cycles of revumenib therapy. Each cycle is 28 days.
Cumulative incidence of infections | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ball, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States